CLINICAL TRIAL: NCT05475288
Title: Incidence, Risk Factor, Treatment and Overall Survival of Locoregionally Recurrent Colon Cancer: a Retrospective, Population-based Cohort Study
Brief Title: Incidence, Risk Factor, Treatment and Overall Survival of Locoregionally Recurrent Colon Cancer
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Hidde Swartjes, Researcher in training, Radboud University Medical Center
Other Study IDs: K20.306
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Colonic Neoplasms; Neoplasm Recurrence, Local
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on disease recurrence was collected for all primary colon cancer patients diagnosed in the Netherlands over the first six months of 2015. Three-year cumulative incidence, risk factors, treatment and three-year OS of locoregionally recurrent colon cancer were determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage I-III primary colon carcinoma;
* Diagnosed between January 1st and June 30th of 2015;
* Surgical resection of primary colon carcinoma.

Exclusion Criteria:

* Appendiceal localization;
* Neuroendocrine tumor morphology;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with stage I-III primary colon cancer in the first half of 2015.
Sampling Method: Non-Probability Sample
Enrollment: 3554 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of patients with locoregionally recurrent colon cancer in curatively treated primary colon cancer patients | Three years
  UNIT OF MEASUREMENT: Cumulative incidence of patients with locoregionally recurrent colon cancer in curatively treated primary colon cancer patients; MEASUREMENT TOOL: Registration of diagnosis of locoregionally recurrent colon cancer in the electronic patient file.
  The competing-risk cumulative incidence will be calculated, which will inform on the proportion of patients who have developed locoregionally recurrent colon cancer at that time point.
Risk factors for development of locoregionally recurrent colon cancer in primary colon cancer patients | Three years
  UNIT OF MEASUREMENT: Risk factors for development of locoregionally recurrent colon cancer in primary colon cancer patients; MEASUREMENT TOOL: Registration of clinical and pathological covariates of primary colon cancer in the electronic patient file and national pathological database (PALGA).
  Clinical and pathological risk factors for the development of locoregionally recurrent colon cancer will be identified using multivariable competing-risk risk regression analyses, according to the cause-specific hazard approach. This will inform on specific clinical and pathological covariates which increase or decrease the risk for development of locoregionally recurrent colon cancer.
Proportions of treatment given to patients with locoregionally recurrent colon cancer | Three years
  UNIT OF MEASUREMENT: Proportions of treatment given to patients with locoregionally recurrent colon cancer; MEASUREMENT TOOL: Registration of treatment for locoregionally recurrent colon cancer in the electronic patient file.
  Using descriptive statistics, treatment patterns of patients with locoregionally recurrent colon cancer will be identified. Groups that will be created, will also be used to assess overall survival.
Overall survival of patients with locoregionally recurrent colon cancer; | Three years
  UNIT OF MEASUREMENT: Overall survival of patients with locoregionally recurrent colon cancer; MEASUREMENT TOOL: Registration of vital status in the national personal records database.
  Overall survival will be estimated for patients with locoregionally recurrent colon cancer, stratifying for different groups (i.e. treatment, diagnosis of synchronous metastases, diagnosis within first year after primary resection, etc.)

IPD SHARING:
Plan to Share IPD: No
Data can be requested through the Netherlands Cancer Registry.

REFERENCES:
- [Derived] Swartjes H, van Lankveld DWP, van Erning FN, Verheul HMW, de Wilt JHW, Koeter T, Vissers PAJ. Locoregionally Recurrent Colon Cancer: How Far Have We Come? A Population-Based, Retrospective Cohort Study. Ann Surg Oncol. 2023 Mar;30(3):1726-1734. doi: 10.1245/s10434-022-12689-5. Epub 2022 Oct 19. PMID 36261752